CLINICAL TRIAL: NCT06201104
Title: The Effect of Patient Empowerment Training on Patients' Self-Efficacy, Health Locus of Control and Perception of Nursing Care Quality
Brief Title: Patient Empowerment Training for COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Filiz Ozbey, Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022/119
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: patient; empowerment education; self-efficacy; health locus of control; quality of nursing care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Two pulmonology services will be selected by lottery among a total of 9 pulmonology services. Among two chest diseases services, patients will be randomly assigned, one in the experimental group and the other in the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The data of the research will be collected by a statistics expert who has no knowledge of the research process. Patients will not know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will be given patient empowerment training as an intervention. The aim of the training is to ensure that patients have the knowledge, skills and attitudes necessary to manage the care and treatment processes both during their hospitalization and in their daily lives after discharge.
  Interventions: Other: Patient empowerment education
- Control group (No Intervention): After the pre-test data is collected from the control group by face-to-face interview method, no intervention will be made to the control group. At the end of the second month, the same scales will be re-administered over the phone as post-test data.

INTERVENTIONS:
Other: Patient empowerment education — After the pre-test is administered to the patients in the experimental group, patient empowerment training (intervention) will be given. Patients will be divided into groups of 15 people and the training will be given in a total of 6 sessions, all in one session. The "Patient Empowerment Handbook" prepared by the researchers will be used during the training. The training was planned to last 1 hour (45 minutes of theoretical training, 15 minutes of question and answer). The training was planned to be carried out in an interactive manner (question and answer method, sharing of patient experiences, group discussion). The "Patient Empowerment Handbook" will be delivered to patients after the training for them to read whenever they want. How to use the manual will be explained to patients.
  Arms: Experimental group

SUMMARY:
The aim of the study, planned in a randomized, pre-test, post-test, control group and single-blind research design, is to examine the effect of empowerment training given to inpatients diagnosed with chronic obstructive pulmonary disease (COPD) on the patients' self-efficacy, health locus of control and perception of nursing care quality. The population of the research will consist of patients (N=6000) diagnosed with chronic obstructive pulmonary disease (COPD) who are receiving inpatient treatment in any two chest diseases services of a training and research hospital (EAH) that provides tertiary healthcare services on the European side of Istanbul. Two pulmonology services will be selected by lottery among a total of 9 pulmonology services. Among two chest diseases services, patients will be randomly assigned, one in the experimental group and the other in the control group. Patients' data will be collected with the Introductory Information Form, COPD Information Survey, Generalized Self-Efficacy Scale, Multidimensional Health Locus of Control Scale Form A and Care Behavior Scale-24. The data of the study will be analyzed using descriptive tests, intergroup comparison tests and correlation analysis.

Key Words: Patient, empowerment education, self-efficacy, health locus of control, nursing care quality.

DETAILED DESCRIPTION:
The aim of the study, planned in a randomized, pre-test, post-test, control group and single-blind research design, is to examine the effect of empowerment training given to inpatients diagnosed with chronic obstructive pulmonary disease (COPD) on the patients' self-efficacy, health locus of control and perception of nursing care quality. In line with the purpose of the research, the hypotheses were determined as follows:

H1-0: Strength training has no effect on patients' self-efficacy. H1-1: Empowerment training has an effect on patients' self-efficacy. H2-0: Strength training has no effect on patients' health locus of control. H2-1: Strength training has an effect on patients' health locus of control. H3-0: Empowerment education has no effect on patients' perception of nursing care quality.

H3-1: Empowerment education has an effect on patients' perception of nursing care quality.

The population of the research will consist of patients (N=6000) diagnosed with chronic obstructive pulmonary disease (COPD) who are receiving inpatient treatment in any two chest diseases services of a training and research hospital (EAH) that provides tertiary healthcare services on the European side of Istanbul. Two pulmonology services will be selected by lottery among a total of 9 pulmonology services. Among two chest diseases services, patients will be randomly assigned, one in the experimental group and the other in the control group. The determination of the experimental and control groups will be carried out in a single blind manner and in a computer environment by an external expert. In the research, provided that the number of patients in the experimental and control groups is equal, the patients will be numbered in the order of admission to the ward (taking into account first the date and then the time) until 182 patients are reached and they will be assigned to the experimental and control groups in a random manner. Preliminary implementation of the study will be carried out before patients are assigned to the experimental and control groups. Permission will be obtained for the preliminary application of the research. 3 COPD patients hospitalized in the chest diseases services of EAH and who agree to participate in the preliminary application will be asked to answer the questions in the data collection tools and read the patient empowerment training brochure. Patients' data will be collected with the Introductory Information Form, COPD Information Survey, Generalized Self-Efficacy Scale, Multidimensional Health Locus of Control Scale Form A and Care Behavior Scale-24. The data of the study will be analyzed using descriptive tests, intergroup comparison tests and correlation analysis.

Key Words: Patient, empowerment education, self-efficacy, health locus of control, nursing care quality.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months have passed since the diagnosis of COPD,
* Having received inpatient treatment in the hospital for at least two nights,
* Being conscious,
* No communication barrier,
* Being literate in Turkish,
* Being 18 years or older,
* Agreeing to participate in the research.

Exclusion Criteria:

* General health condition is not suitable to participate in the training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in patients' self-efficacy after education | Two months
  Scales
Change in patients' health locus of control after education | Two months
  Scales
Change in patients' perception of nursing care quality after education | Two months
  Scales

CONTACTS AND LOCATIONS:
Overall Officials: Betül Sönmez, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)